CLINICAL TRIAL: NCT02008721
Title: Double-blind, Randomised, Placebo-controlled Parallel Group Study to Investigate the Effect of EGCG Supplementation on Disease Progression of Patients With Multiple System Atrophy (MSA)
Brief Title: Progression Rate of MSA Under EGCG Supplementation as Anti-Aggregation-Approach
Acronym: PROMESA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Johannes Levin (Other)
Collaborators: German Center for Neurodegenerative Diseases (DZNE) (Other); Deutsche Parkinson Vereinigung (Other); German Foundation for Neurology (Other); ParkinsonFonds Deutschland gGmbH (Other)
Responsible Party: Sponsor-Investigator, Dr. Johannes Levin, Sponsor delegated person, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PROMESA
Record Dates: First submitted 2013-12-08; First posted 2013-12-11 (Estimated); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-08

CONDITIONS: Multiple System Atrophy
Keywords: Multiple System Atrophy; epigallocatechin gallate
MeSH Terms: conditions — Multiple System Atrophy | interventions — epigallocatechin gallate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EGCG as putative neuroprotective agent (Active Comparator): Treatment with 800 mg - 1200 mg EGCG as putative neuroprotective agent
  Interventions: Drug: EGCG as putative neuroprotective agent
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EGCG as putative neuroprotective agent — Treatment with 800 mg - 1200 mg EGCG as putative neuroprotective agent
  Other Names: Sunphenon EGCg
  Arms: EGCG as putative neuroprotective agent
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
MSA is a rapidly progressive disorder with an average survival time of about 7 years after the first clinical manifestation. No potent symptomatic treatment is currently available. A disease-modifying therapy does not exist either. The growing understanding in recent years of the underlying pathological mechanisms of the disease allows the development of new treatment options that have a modifying effect on the disease progression. Therefore, treatments are urgently required that effect the central underlying pathological mechanism, which appears to be the intracellular aggregation of toxic oligomers of α-synuclein.

EGCG, a polyphenol found in green tea, has shown to inhibit the formation of toxic α-synuclein oligomers in vitro and has shown to transform α-synuclein-oligomers in non-toxic oligomer species. There is also evidence for a neuroprotective effect in MPTP-mouse models of PD and is an antioxidant and iron chelator. There are currently 63 clinical studies (http://clinicaltrial.gov) in which EGCG was applied for various indications, such as Multiple Sclerosis, various forms of cancer and Huntington's disease. All of which have shown good tolerability and safety with the applied doses of EGCG of up to 1200 mg per day, demonstrating the safety of the drug under controlled clinical conditions (see 5.3.1 for hepatotoxicity in uncontrolled conditions).

These data provide a solid rationale for testing in a clinical trial if supplementation of EGCG can interfere with the core disease mechanism in MSA and consequently retard the clinical progression of the MSA-related disability.

DETAILED DESCRIPTION:
5 Introduction Multiple System Atrophy (MSA) is a slowly progressing neurodegenerative disease that is characterized by i) a hypokinetic movement disorder which defines MSA of the parkinsonian type (MSA-P) or by ii) cerebellar symptoms which define MSA of the cerebellar type (MSA-C). In both types the movement disorder can be accompanied by vegetative symptoms such as orthostatic hypotension. In contrast to Parkinson's disease (PD), the effect of dopaminergic medication on the parkinsonian symptoms is very limited. In spite of several efforts, no disease modifying therapy has been identified so far. Several lines of evidence including epidemiological, in vitro, and in vivo data, suggest that Epigallocatechin gallate (EGCG) might be able to delay disease progression of MSA by modifying several aspects in the pathogenesis of MSA such as protein aggregation, oxidative stress and iron accumulation. Therefore, this study is designed to investigate the influence of EGCG on disease progression in patients with MSA. To assess the effect on disease progression, clinical evaluation and MR-imaging will be applied in a bi-center, prospective, placebo-controlled, double-blind randomized phase III trial. The primary outcome measure will be the change in motor symptoms from V1 to V7 measured by the UMSARS-ME comparing placebo- vs. verum-treated patients. The secondary efficacy endpoint will be the change from V1 to V7 in the total UMSARS score, in the CGI score and in MRI parameters (global and regional atrophy / iron deposition) comparing placebo- vs. verum-treated patients.

5.1 Background The disease: MSA is a synucleinopathy that is suitable for various reasons as a model disease to investigate disease-modifying effects in α-synuclein (aSyn)-dependent neurodegeneration. The disease progression is more rapid compared to PD and therefore allows the observation of clinically relevant effects in shorter observation periods. As no potent symptomatic treatment of MSA is currently available, the influence of symptomatic active substances on clinical data is limited and placebo can be used as comparator. This solves the potential ethical problem of having to deprive patients of such symptomatic treatment during the study and underlines the high medical need for a symptomatic treatment. Another important argument for neuroprotection studies in MSA is that in three independent studies EMSA, NNIPPS, MEMSA a very similar disease progression was observed over a defined period of time, which enables a precise power analysis with sample sizes and follow-up periods that are suitable for an investigator initiated trial (IIT).

The therapeutic target: An increasing amount of data suggests that toxic oligomers from misfolded, disease-specific proteins play a potentially important role in the neuronal cell death in neurodegenerative diseases. Specifically in MSA, oligomeric aSyn aggregate species appear to be crucially involved in the pathogenetic mechanisms.

The pharmacological compound: Epidemiological data suggest that ingredients in tea may be neuroprotective for synucleinopathies in man. Regular consumption of tea reduces the risk of contracting PD by about 50%. Also for MSA, a clear trend in the sense of a positive effect of tea consumption on the risk of disease development was observed (OR = 0.5, 95% CI: 0.22-1.5, p = 0.09). EGCG, a polyphenol that is for example found in green tea, inhibits the formation of toxic aSyn oligomers in vitro and transforms aSyn oligomers by direct interaction in alternative, non-toxic oligomer species. Furthermore, EGCG shows a neuroprotective effect in the 1-Methyl-4-phenyl-1,2,3,6-tetrahydropyridin (MPTP) mouse model of PD. In addition, EGCG is an antioxidant and an iron chelator and therefore has more potential beneficial effects on synucleinopathies.

The pharmacokinetic properties of EGCG were tested in humans in the serum and in rodents in serum and organs, including the brain in detail. It was found that repeated oral application of doses of EGCG result in a significant increase in serum levels in healthy adults compared to a single dose. The proposed daily dose of 1200 mg of EGCG is comparable to about 15 to 30 cups of green tea (depending on the mode of preparation) (Prof. F. Paul, Berlin, pers. comm.). Animal experiments in rodents have shown that after a single i.v. dose of EGCG, the substance is found in the brain in significant quantities.

5.2 Trial Rationale MSA is a rapidly progressive disorder with an average survival time of about 7 years after the first clinical manifestation. No potent symptomatic treatment is currently available. A disease-modifying therapy does not exist either. The growing understanding in recent years of the underlying pathological mechanisms of the disease allows the development of new treatment options that have a modifying effect on the disease progression. Therefore, treatments are urgently required that effect the central underlying pathological mechanism, which appears to be the intracellular aggregation of toxic oligomers of aSyn.

EGCG, a polyphenol found in green tea, has shown to inhibit the formation of toxic aSyn oligomers in vitro and has shown to transform aSyn-oligomers in non-toxic oligomer species. There is also evidence for a neuroprotective effect in MPTP-mouse models of PD and is an antioxidant and iron chelator. There are currently 63 clinical studies in which EGCG was applied for various indications, such as Multiple Sclerosis, various forms of cancer and Huntington's disease. All of which have shown good tolerability and safety with the applied doses of EGCG of up to 1200 mg per day, demonstrating the safety of the drug under controlled clinical conditions.

These data provide a solid rationale for testing in a clinical trial if supplementation of EGCG can interfere with the core disease mechanism in MSA and consequently retard the clinical progression of the MSA-related disability.

5.3 Side effects and Risk Benefit Assessment 5.3.1 Side effects In all clinical trials investigating the oral intake of green tea/EGCG in various doses and pharmacological forms, EGCG has shown a good safety and tolerability in daily doses of up to 1200 mg over a period of 6 months. Side effects that have been reported after application of EGCG were usually mild and did not occur more often than under placebo (flatulence, headache, nausea, vertigo, abdominal cramps and muscle pain). Other reported side effects (arterial hypertension, palpitations, headache, polyuria, tremor, sleep disorders, nausea/vomiting) are due to the caffeine part in green tea and are not due to EGCG, as all studies using pure EGCG have not reported such side effects.

No relevant or persistent changes in the extensive clinical serum tests have been found so far; also no influence on vital parameters have been reported after using EGCG. Only minimal and transient changes of the blood pressure, echocardiography, liver function tests and serum lipids have been reported. In a study of Chow et al. healthy subjects were given 800 mg EGCG or Polyphenon E (a mixture of several green tea extracts with a 50-75%share of EGCG) once daily or 400 mg twice daily versus placebo over a period of 4 weeks. Only mild side effects occurred in several subjects (flatulence, abdominal pain, nausea, headache, dizziness and muscle pain) that were not occurring more often than under placebo.

The SuniMS study, NCT ID: 00525668, recorded no SUSAR in 120 patients with remitting-relapsing MS, who were administered 800 mg Sunphenon/ EGCG per day. They also were able to show an excellent tolerability. Only 15 patients showed mild, clinically insignificant elevations of liver function tests, which are not necessarily caused by the study medication. The ongoing SUPREMES study, NCT ID: 00799, has so far not recorded any SUSAR in 60 patients with progressive MS who have been on up to 1200 mg EGCG/day for up to 48 months.

In a study by Chen et al a significant protective effect of orally applied EGCG could be demonstrated in mice with a toxic liver failure caused by tetrachlorohydrocarbons. Otherwise, single cases of hepatotoxicity following application of various forms of green tea polyphenols are known. In the period between 1999 and 2008, 34 such case reports have been published, 29 of which have shown a positive de-challenge and 7 have shown a positive re-challenge. The clinical and pathological symptoms included mild elevations of liver function tests, cholestasis, cholangitis, hepatocellular inflammation and hepatocellular necrosis. The symptoms were usually completely reversible after stopping the medication. One patient died of liver failure. Signs of liver toxicity were recorded between day 9 up to 5 months after beginning a therapy with doses of 187,5 -468,75mg EGCG/day).

The withdrawal of a green tea extract in Spain and France (Exolise®) a couple of years ago needs to be mentioned. After application of this medication some cases of severe hepatotoxicity were reported. Symptoms like icterus, massive elevation of transaminases occurred not later than 12 weeks after beginning the treatment with the extract in capsules and were completely reversible few weeks after stopping the medication. The exact underlying mechanisms have not been completely worked out. Possibly these are due to a SAE that is specific for Exolise®, and is connected with the manufacturing process (hydro-alcoholic extraction techniques). For this reason, only the distribution of Exolise® has been stopped by the respective authorities, but not the distribution of other green tea extracts (see also the following publications by the WHO): www.who.int/entity/medicines/publications/restrictedpharm2005.pdf It has not yet been found out which parts of the polyphenols and their metabolites are responsible for the hepatotoxic effects. Even though in most cases mixtures of green tea and polyphenols have been administered it is suspected, that EGCG as a main component of the green tea extracts shows hepatotoxic potential. In favor of this hypothesis is the fact, that there have been reports of elevated transaminases under treatment with EGCG in man and interactions with other substances. EGCG is known to bind to α- and β-estrogene receptors and increases 17 β-estradiol-induced reactions in mice. EGCG is a known inhibitor of the Catechol-O-methyltransferase (COMT) that catalyses the degradation of exogenous and endogenous substances.

It is suspected, that for the biotransformation of green tea catechines, COMT plays an important role. COMT polymorphisms with low activity of COMT could result in elevated plasma levels of toxic EGCG metabolites.

The cytotoxicity of EGCG in hepatocytes seems to be low in vitro and only doses that are higher by a multiple compared to the doses used in clinical studies lead to liver necrosis in animal models. Also, the extremely low bioavailability in man has to be considered.

On the basis of all recent studies using green tea extract and EGCG there are no reports of persistent and severe influence on the physiological systems (blood circulation, respiratory system, central nervous system and urinary tract). Still there are singular case reports of hepatotoxic effects in the context of intake of green tea extracts/ EGCG.

As a conclusion, all data are in favor of a good tolerability of the substance. For further details see the investigator's brochure (Polyphenon E).

5.3.2 Risk Benefit Assessment The reported data suggest a safe pharmacological profile apart from individual cases of hepatotoxicity which can be controlled for by routine serum liver parameters. The preclinical data suggest a molecular mode of action for EGCG which appears to target core pathological mechanisms active in MSA. In absence of any effective symptomatic, protective or curative intervention in this devastating disorder, the risk benefit evaluation justifies the conduct of the proposed clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. "clinical possible" or "clinical probable" MSA (Gilman et al., Neurology, 2008 26;71:670-6)
2. Hoehn & Yahr stage I - III
3. A stable regimen for at least 1 month prior to V1 and willingness / no fore-seeable need to change the regimen throughout the 52 week follow-up pe-riod for

   1. drugs acting against Parkinsonism (e.g. Levodopa, Dopamine-Agonists, Amantadine and MAO-B-Inhibitors)
   2. drugs acting against autonomic dysfunction (e.g. ephedrin, midodrin, fludrucortison, octreotide, desmopresin, oxybutinine)
   3. antidepressant and antidementive drugs.
4. No regular consumption of EGCG, green tea, or more than two cups of black tea per day
5. Capability and willingness to give written informed consent indicating that the subject has been informed of and understood all aspects pertinent to the study
6. Capability and willingness to comply with the procedures of the study
7. Contraception by adequate contraceptive methods (oral, injected or im-planted hormonal contraceptive methods, intrauterine pessar, sterilisation or real abstinence) in all female patients with childbearing potential
8. Absence of liver disease documented by transaminases and bilirubin below 2-folds of the upper normal level.

Exclusion Criteria:

1. Hoehn & Yahr stage > III (loss of postural reflexes, no independent walking possible, inability to stand unassisted, wheelchair-bound).
2. Neurodegenerative diseases other than MSA
3. Severe liver disease with elevation of transaminases and bilirubin above 2-folds of the upper normal level or regular intake of hepatotoxic drugs
4. Known hypersensitivity to EGCG or to drugs with similar chemical structure
5. Participation in another clinical trial involving administration of an investigational medicinal product within 1 month prior to V1
6. A physical or psychiatric condition, which at the investigator's discretion may put the subject at risk, may confound the trial results, or may interfere with the subject's participation in this clinical trial
7. Persistent abuse of medication, drugs or alcohol
8. Consumption of > 500 ml grapefruit juice per day (leading to inhibition of cytochrome P-450 isoenzyme 3A4, which may be involved in degradation of EGCG).
9. Current or planned pregnancy or breast feeding in females
10. Females of childbearing potential, who are not using medically reliable methods of contraception for the entire study duration (such as oral, inject-able, or implantable contraceptives, or intrauterine contraceptive devices).
11. Intake of COMT-inhibitors (e.g. Entacapone, Tolcapone)
12. Current or planned therapy with Bortezomib and/ or history of plasmocytoma.
13. Anemia at Screening (Hb < 10g/dl)
14. Other severe medical conditions upon discretion of the LKP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2014-01; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Levin, MD, Principal Investigator — Ludwig Maximilians University, Department of Neurology; Günter Höglinger, MD, Principal Investigator — Deutsches Zentrum für Neurodegenerative Erkrankungen e.V.
Locations (12):
- Germany (12):
  - Neurology Department, Ludwig-Maximilians University, München, Bavaria
  - Department of Neurology, Klinikum rechts der Isar, Technische Universität München, München, Bavaria
  - Kliniken Beelitz GmbH, Neurologisches Fachkrankenhaus für Bewegungsstörungen, Beelitz-Heilstätten
  - Charité - Universitätsmedizin Berlin, Berlin
  - Technische Universität Dresden, Dresden
  - Heinrich-Heine-Universität, Neurologische Klinik, Düsseldorf
  - Paracelsus-Elena-Klinik Kassel, Kassel
  - Universität Leipzig, Leipzig
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Philipps Universität Marburg, Marburg
  - Eberhard Karls Universität Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm

REFERENCES:
- [Background] Gilman S, Wenning GK, Low PA, Brooks DJ, Mathias CJ, Trojanowski JQ, Wood NW, Colosimo C, Durr A, Fowler CJ, Kaufmann H, Klockgether T, Lees A, Poewe W, Quinn N, Revesz T, Robertson D, Sandroni P, Seppi K, Vidailhet M. Second consensus statement on the diagnosis of multiple system atrophy. Neurology. 2008 Aug 26;71(9):670-6. doi: 10.1212/01.wnl.0000324625.00404.15. PMID 18725592
- [Background] Wenning GK, Tison F, Seppi K, Sampaio C, Diem A, Yekhlef F, Ghorayeb I, Ory F, Galitzky M, Scaravilli T, Bozi M, Colosimo C, Gilman S, Shults CW, Quinn NP, Rascol O, Poewe W; Multiple System Atrophy Study Group. Development and validation of the Unified Multiple System Atrophy Rating Scale (UMSARS). Mov Disord. 2004 Dec;19(12):1391-402. doi: 10.1002/mds.20255. PMID 15452868
- [Background] Dodel R, Spottke A, Gerhard A, Reuss A, Reinecker S, Schimke N, Trenkwalder C, Sixel-Doring F, Herting B, Kamm C, Gasser T, Sawires M, Geser F, Kollensperger M, Seppi K, Kloss M, Krause M, Daniels C, Deuschl G, Bottger S, Naumann M, Lipp A, Gruber D, Kupsch A, Du Y, Turkheimer F, Brooks DJ, Klockgether T, Poewe W, Wenning G, Schade-Brittinger C, Oertel WH, Eggert K. Minocycline 1-year therapy in multiple-system-atrophy: effect on clinical symptoms and [(11)C] (R)-PK11195 PET (MEMSA-trial). Mov Disord. 2010 Jan 15;25(1):97-107. doi: 10.1002/mds.22732. PMID 20014118
- [Background] Kragh CL, Lund LB, Febbraro F, Hansen HD, Gai WP, El-Agnaf O, Richter-Landsberg C, Jensen PH. Alpha-synuclein aggregation and Ser-129 phosphorylation-dependent cell death in oligodendroglial cells. J Biol Chem. 2009 Apr 10;284(15):10211-22. doi: 10.1074/jbc.M809671200. Epub 2009 Feb 9. PMID 19203998
- [Background] Checkoway H, Powers K, Smith-Weller T, Franklin GM, Longstreth WT Jr, Swanson PD. Parkinson's disease risks associated with cigarette smoking, alcohol consumption, and caffeine intake. Am J Epidemiol. 2002 Apr 15;155(8):732-8. doi: 10.1093/aje/155.8.732. PMID 11943691
- [Background] Tan EK, Tan C, Fook-Chong SM, Lum SY, Chai A, Chung H, Shen H, Zhao Y, Teoh ML, Yih Y, Pavanni R, Chandran VR, Wong MC. Dose-dependent protective effect of coffee, tea, and smoking in Parkinson's disease: a study in ethnic Chinese. J Neurol Sci. 2003 Dec 15;216(1):163-7. doi: 10.1016/j.jns.2003.07.006. PMID 14607318
- [Background] Vidal JS, Vidailhet M, Elbaz A, Derkinderen P, Tzourio C, Alperovitch A. Risk factors of multiple system atrophy: a case-control study in French patients. Mov Disord. 2008 Apr 30;23(6):797-803. doi: 10.1002/mds.21857. PMID 18307243
- [Background] Bieschke J, Russ J, Friedrich RP, Ehrnhoefer DE, Wobst H, Neugebauer K, Wanker EE. EGCG remodels mature alpha-synuclein and amyloid-beta fibrils and reduces cellular toxicity. Proc Natl Acad Sci U S A. 2010 Apr 27;107(17):7710-5. doi: 10.1073/pnas.0910723107. Epub 2010 Apr 12. PMID 20385841
- [Background] Levites Y, Weinreb O, Maor G, Youdim MB, Mandel S. Green tea polyphenol (-)-epigallocatechin-3-gallate prevents N-methyl-4-phenyl-1,2,3,6-tetrahydropyridine-induced dopaminergic neurodegeneration. J Neurochem. 2001 Sep;78(5):1073-82. doi: 10.1046/j.1471-4159.2001.00490.x. PMID 11553681
- [Background] Ullmann U, Haller J, Decourt JD, Girault J, Spitzer V, Weber P. Plasma-kinetic characteristics of purified and isolated green tea catechin epigallocatechin gallate (EGCG) after 10 days repeated dosing in healthy volunteers. Int J Vitam Nutr Res. 2004 Jul;74(4):269-78. doi: 10.1024/0300-9831.74.4.269. PMID 15580809
- [Background] Lin LC, Wang MN, Tseng TY, Sung JS, Tsai TH. Pharmacokinetics of (-)-epigallocatechin-3-gallate in conscious and freely moving rats and its brain regional distribution. J Agric Food Chem. 2007 Feb 21;55(4):1517-24. doi: 10.1021/jf062816a. Epub 2007 Jan 27. PMID 17256961
- [Background] Chow HH, Cai Y, Hakim IA, Crowell JA, Shahi F, Brooks CA, Dorr RT, Hara Y, Alberts DS. Pharmacokinetics and safety of green tea polyphenols after multiple-dose administration of epigallocatechin gallate and polyphenon E in healthy individuals. Clin Cancer Res. 2003 Aug 15;9(9):3312-9. PMID 12960117
- [Background] Bettuzzi S, Brausi M, Rizzi F, Castagnetti G, Peracchia G, Corti A. Chemoprevention of human prostate cancer by oral administration of green tea catechins in volunteers with high-grade prostate intraepithelial neoplasia: a preliminary report from a one-year proof-of-principle study. Cancer Res. 2006 Jan 15;66(2):1234-40. doi: 10.1158/0008-5472.CAN-05-1145. PMID 16424063
- [Background] Wang Y, Butros SR, Shuai X, Dai Y, Chen C, Liu M, Haacke EM, Hu J, Xu H. Different iron-deposition patterns of multiple system atrophy with predominant parkinsonism and idiopathetic Parkinson diseases demonstrated by phase-corrected susceptibility-weighted imaging. AJNR Am J Neuroradiol. 2012 Feb;33(2):266-73. doi: 10.3174/ajnr.A2765. Epub 2011 Nov 3. PMID 22051807
- [Background] Huppertz HJ, Kroll-Seger J, Kloppel S, Ganz RE, Kassubek J. Intra- and interscanner variability of automated voxel-based volumetry based on a 3D probabilistic atlas of human cerebral structures. Neuroimage. 2010 Feb 1;49(3):2216-24. doi: 10.1016/j.neuroimage.2009.10.066. Epub 2009 Oct 28. PMID 19878722
- [Background] Schweser F, Sommer K, Deistung A, Reichenbach JR. Quantitative susceptibility mapping for investigating subtle susceptibility variations in the human brain. Neuroimage. 2012 Sep;62(3):2083-100. doi: 10.1016/j.neuroimage.2012.05.067. Epub 2012 Jun 1. PMID 22659482
- [Background] Schweser F, Deistung A, Lehr BW, Reichenbach JR. Differentiation between diamagnetic and paramagnetic cerebral lesions based on magnetic susceptibility mapping. Med Phys. 2010 Oct;37(10):5165-78. doi: 10.1118/1.3481505. PMID 21089750
- [Background] Caruana M, Hogen T, Levin J, Hillmer A, Giese A, Vassallo N. Inhibition and disaggregation of alpha-synuclein oligomers by natural polyphenolic compounds. FEBS Lett. 2011 Apr 20;585(8):1113-20. doi: 10.1016/j.febslet.2011.03.046. Epub 2011 Mar 31. PMID 21443877
- [Derived] Levin J, Maass S, Schuberth M, Giese A, Oertel WH, Poewe W, Trenkwalder C, Wenning GK, Mansmann U, Sudmeyer M, Eggert K, Mollenhauer B, Lipp A, Lohle M, Classen J, Munchau A, Kassubek J, Gandor F, Berg D, Egert-Schwender S, Eberhardt C, Paul F, Botzel K, Ertl-Wagner B, Huppertz HJ, Ricard I, Hoglinger GU; PROMESA Study Group. Safety and efficacy of epigallocatechin gallate in multiple system atrophy (PROMESA): a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2019 Aug;18(8):724-735. doi: 10.1016/S1474-4422(19)30141-3. Epub 2019 Jul 2. PMID 31278067
- See also: Fox trial finder of the Michael J Fox foundation — http://foxtrialfinder.michaeljfox.org/pages/find-trials/default.aspx/?keywords=PROMESA

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EGCG as Putative Neuroprotective Agent | Placebo
Started | 47 | 45
Completion of Study Assessment | 31 | 33
Completion Without Protocol Violation | 30 | 33
Participation in MRI Substudy | 17 | 15
Completion of MRI Substudy | 11 | 8
Completed | 32 | 35
Not Completed | 15 | 10
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Death | 4 | 2
Not completed — Adverse Event | 3 | 5
Not completed — Protocol Violation | 3 | 2

BASELINE CHARACTERISTICS:
Population: Patients with both, the parkinsonian (MSA-P) and cerebellar variant of MSA (MSA-C) respectively were included. At screening, participants had to be able to ambulate independently and to abstain from regular consumption of EGCG, green tea or more than two cups of black tea per day.
Groups:
- Total: Total of all reporting groups
Arm/Group | EGCG as Putative Neuroprotective Agent | Placebo | Total
Number analyzed (Participants) | 47 | 45 | 92
Age, Continuous [Median (Full Range); unit: years] | 60 [56 to 71] | 64 [60 to 70] | 62 [56 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 29 | 26 | 55
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 47 | 45 | 92

OUTCOME MEASURES:

1. Primary Outcome: Change of Score in Motor Examination (ME) of the Unified MSA Rating Scale (UMSARS-ME) From V1 to V7.
Description: To assess the efficacy of EGCG vs. Placebo to reduce the progression in the motor examination (ME) of the Unified MSA Rating Scale (UMSARS-ME) from V1 to V7.
  The UMSARS-ME (Unified Multiple System Atrophy Rating Scale, Motor examination) assesses 14 operationalised signs of multiple system atrophy. 25 Scores for all 14 items range from 0 to 4, thus total scores range from 0 to 56. Higher scores mean a worse outcome.
Time Frame: 52 weeks
Population: Eligible patients were older than 30 years; met the diagnostic criteria for possible or probable parkinsonism-predominant or cerebellar-ataxia-predominant multiple system atrophy; could ambulate independently (ie, Hoehn and Yahr stages 1-3); and had to be on stable anti-Parkinson's, anti-dysautonomia, anti-dementia, and anti-depressant regimens.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EGCG as Putative Neuroprotective Agent | Placebo
Number analyzed (Participants) | 47 | 45
score on a scale | 5.66 (1.01) | 6.60 (0.99)
Statistical Analysis 1: Comparison: EGCG as Putative Neuroprotective Agent vs Placebo; Power calculation: 80% power, 5% P-level, 50% effect size, i.e. an expected mean yearly UMSARS-ME increase of 3,9 under verum treatment compared to 7.8 ± 6.8 (mean ± standard deviation) under Placebo treatment. We used a linear mixed-effects model to test the primary hypothesis-ie, to compare differences in the change in motor examination scores on UMSARS between baseline and week 52 between the study groups; Test type: Superiority; p = 0.51, Mixed Models Analysis

2. Secondary Outcome: Possible Symptomatic Effects of EGCG vs. Placebo Measured by the Change in the UMSARS - ME in the Wash-out Phase (From V6-V7)
Description: To assess any effect of EGCG vs. Placebo on the evolution of the above mentioned parameters during the wash-out phase (from V6-V7) measured by the UMSARS - ME.
  The UMSARS-ME (Unified Multiple System Atrophy Rating Scale, Motor examination) assesses 14 operationalised signs of multiple system atrophy. 25 Scores for all 14 items range from 0 to 4, thus total scores range from 0 to 56. Higher scores mean a worse outcome.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EGCG as Putative Neuroprotective Agent | Placebo
Number analyzed (Participants) | 47 | 45
score on a scale | 0.68 (0.60) | 0.49 (0.58)
Statistical Analysis 1: Comparison: EGCG as Putative Neuroprotective Agent vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.82, Mixed Models Analysis

3. Secondary Outcome: Change in the UMSARS Total Score From V1 to V7
Description: To assess the efficacy of EGCG vs. Placebo to reduce the progression from V1 to V7 in UMSARS total score
  The total score of the UMSARS (Unified Multiple System Atrophy Rating Scale) is a disease specific rating scale that comprises the activities of daily living subscale and the motor examination subscale.
  The activities of daily living subscale assesses motor symptoms and autonomic symptoms (items 1-12 of the UMSARS activities of daily living subscale) with scores from 0-4 for every item, resulting in a minimum score of 0 and a maximum score of 48. A higher score means a worse outcome. It also includes the 14 items of the UMSARS motor examination subscale with possible scores from 0-4 for every item, resulting in a score range from 0-56. The UMSARS total score hence shows a range from 0 to 104.
  Higher scores indicate a greater impairment.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EGCG as Putative Neuroprotective Agent | Placebo
Number analyzed (Participants) | 47 | 45
score on a scale | 10.33 (1.73) | 10.35 (1.71)
Statistical Analysis 1: Comparison: EGCG as Putative Neuroprotective Agent vs Placebo; Power calculation: 80% power, 5% P-level, 50% effect size. We used a linear mixed-effects model to test the primary hypothesis-ie, to compare differences in the change in UMSARS total score between baseline and week 52 between the study groups. We did a post-hoc power calculation based on the mean change in motor examination scores on UMSARS and SDs in the placebo group of the per-protocol study completer set to test the assumptions of our initial power calculation; Test type: Superiority; p = 0.99, Mixed Models Analysis

4. Secondary Outcome: Possible Symptomatic Effects of EGCG vs. Placebo Measured by the UMSARS Total Score From V6 to V7 (During the Washout Phase)
Description: To assess any effect of EGCG vs. Placebo on the UMSARS total score during the wash-out phase (from V6 to V7) to explore possible symptomatic effects.
  The total score of the UMSARS (Unified Multiple System Atrophy Rating Scale) is a disease specific rating scale that comprises the activities of daily living subscale and the motor examination subscale.
  The activities of daily living subscale assesses motor symptoms and autonomic symptoms (items 1-12 of the UMSARS activities of daily living subscale) with scores from 0-4 for every item, resulting in a minimum score of 0 and a maximum score of 48. A higher score means a worse outcome. It also includes the 14 items of the UMSARS motor examination subscale with possible scores from 0-4 for every item, resulting in a score range from 0-56. The UMSARS total score hence shows a range from 0 to 104, a higher score indicates greater impairment.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EGCG as Putative Neuroprotective Agent | Placebo
Number analyzed (Participants) | 47 | 45
score on a scale | 0.70 (0.91) | -0.29 (0.88)
Statistical Analysis 1: Comparison: EGCG as Putative Neuroprotective Agent vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.43, Mixed Models Analysis

5. Secondary Outcome: Percentage of Striatal Volume Loss in MRI (3D MP-RAGE MRI Volumetry, 3D FLAIR) From Baseline to V7 as Effect of Treatment (Epigallocatechin Gallate vs Placebo)
Description: To assess the efficacy of EGCG vs. Placebo to reduce the progression from V1 to V7 (52 weeks) in striatal volume loss measured by MRI (3D MP-RAGE MRI volumetry, 3D FLAIR)
Time Frame: baseline to 52 weeks
Population: 17 patients in the EGCG-group and 15 patients in the placebo group took part in the MRI substudy.
  A reduced number of 11 patients were analysed in the EGCG group and 8 patients in the Placebo group, as only these patients had taken part in the follow-up MRI assessments.
Measure: Mean (Standard Deviation); unit: % of volume loss
Arm/Group | EGCG as Putative Neuroprotective Agent | Placebo
Number analyzed (Participants) | 11 | 8
% of volume loss | -0.029 (0.027) | -0.064 (0.026)

6. Secondary Outcome: Clinical Safety and Tolerability of EGCG Measured by Death Rates
Description: Clinical safety and tolerability of EGCG measured by number of deaths in EGCG- Group vs Placebo-Group
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | EGCG as Putative Neuroprotective Agent | Placebo
Number analyzed (Participants) | 47 | 45
Participants | 4 | 2

7. Secondary Outcome: Effect of Treatment (Epigallocatechin Gallate vs Placebo) on Safety and Tolerability: Discontinuation Rates Because of Hepatotoxicity
Description: Effect of Treatment (Epigallocatechin Gallate vs Placebo) on Safety and Tolerability: Measured by Discontinuation rates because of hepatotoxicity (measured by increased aminotransferase concentrations)
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | EGCG as Putative Neuroprotective Agent | Placebo
Number analyzed (Participants) | 47 | 45
Participants | 2 | 0

8. Secondary Outcome: Number of Participants Achieving Each Clinical Global Impression of Severity (CGI-S): Illness Level at Visit 1
Description: Clinical Global Impression of Severity (CGI-S) is a 7 item scale that requires the clinician to rate the severity of the patient's illness at the time of assessment.
  Possible ratings are:
  1. Normal, not at all ill
  2. Borderline mentally ill
  3. Mildly ill
  4. Moderately ill
  5. Markedly ill
  6. Severely ill
  7. Among the most extremely ill patients
Time Frame: At baseline visit (max. 4 weeks after the screening visit)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | EGCG as Putative Neuroprotective Agent | Placebo
Number analyzed (Participants) | 47 | 45
participants
  Severity of illness=1 | 2 | 1
  severity of illness =2 | 1 | 0
  severity of illness=3 | 8 | 6
  severity of illness=4 | 23 | 17
  severity of illness=5 | 13 | 20
  severity of illness=6 | 0 | 1
  severity of illness=7 | 0 | 0

9. Secondary Outcome: Number of Participants Achieving Each Clinical Global Impression of Severity (CGI-S): Illness Level at Visit 5
Description: as for outcome 8
Time Frame: Visit 5 (30 weeks after Baseline Visit)
Population: Eligible patients were older than 30 years; met the diagnostic criteria for possible or probable parkinsonism-predominant or cerebellar-ataxia-predominant multiple system atrophy; could ambulate independently (ie, Hoehn and Yahr stages 1-3); and had to be on stable anti-Parkinson's, anti-dysautonomia, anti-dementia, and anti-depressant regimens.
  In the EGCG group only 36 of 47 patients provided data at visit 5 due to SAE/drop out; likewise in the placebo group only 37 of 45 patients.
Measure: Number; unit: participants
Arm/Group | EGCG as Putative Neuroprotective Agent | Placebo
Number analyzed (Participants) | 36 | 37
participants
  Illness Level =1 | 1 | 0
  Illness Level=2 | 1 | 0
  Illness Level =3 | 6 | 5
  Illness Level =4 | 7 | 9
  Illness Level =5 | 15 | 17
  Illness Level =6 | 6 | 6
  Illness Level=7 | 0 | 0

10. Secondary Outcome: Number of Participants Achieving Each Clinical Global Impression of Severity (CGI-S): Illness Level at Visit 6
Description: as for outcome 8
Time Frame: 48 weeks after baseline visit
Population: Eligible patients were older than 30 years; met the diagnostic criteria for possible or probable parkinsonism-predominant or cerebellar-ataxia-predominant multiple system atrophy; could ambulate independently (ie, Hoehn and Yahr stages 1-3); and had to be on stable anti-Parkinson's, anti-dysautonomia, anti-dementia, and anti-depressant regimens.
  In the EGCG group only 32 of 47 patients provided data at visit 6 due to SAE/drop out; likewise in the placebo group only 35 of 45 patients.
Measure: Number; unit: participants
Arm/Group | EGCG as Putative Neuroprotective Agent | Placebo
Number analyzed (Participants) | 32 | 35
participants
  severity of illness=1 | 1 | 0
  severity of illness=2 | 1 | 0
  severity of illness=3 | 6 | 3
  severity of illness=4 | 6 | 12
  severity of illness=5 | 9 | 11
  severity of illness=6 | 9 | 9
  severity of illness=7 | 0 | 0

11. Secondary Outcome: Number of Participants Achieving Each Clinical Global Impression of Severity (CGI-S): Illness Level at Visit 7
Description: Clinical Global Impression of Severity (CGI-S) is a 7 item scale that requires the clinician to rate the severity of the patient's illness at the time of assessment..
  Possible ratings are:
  1. Normal, not at all ill
  2. Borderline mentally ill
  3. Mildly ill
  4. Moderately ill
  5. Markedly ill
  6. Severely ill
  7. Among the most extremely ill patients
Time Frame: 52 weeks after baseline visit
Population: Eligible patients were older than 30 years; met the diagnostic criteria for possible or probable parkinsonism-predominant or cerebellar-ataxia-predominant multiple system atrophy; could ambulate independently (ie, Hoehn and Yahr stages 1-3); and had to be on stable anti-Parkinson's, anti-dysautonomia, anti-dementia, and anti-depressant regimens.
  In the EGCG group only 23 of 47 patients provided data at visit 7 due to SAE/drop out; likewise in the placebo group only 37 of 45 patients.
Measure: Number; unit: participants
Arm/Group | EGCG as Putative Neuroprotective Agent | Placebo
Number analyzed (Participants) | 23 | 37
participants
  severity of illness=1 | 0 | 0
  severity of illness=2 | 1 | 0
  severity of illness=3 | 2 | 3
  severity of illness=4 | 7 | 9
  severity of illness=5 | 9 | 16
  severity of illness=6 | 4 | 8
  severity of illness=7 | 0 | 1

12. Secondary Outcome: Number of Participants Achieving Each Clinical Global Impression of Improvement (CGI-I): Improvement Level at Visit 7 Compared to the Baseline Visit
Description: The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. Compared to the patient's condition at baseline, this patient's condition has either improved or worsened or is unchanged, with a lower score meaning more improvement and a higher score less improvement or worsening respectively. The patient´s state compared to baseline is rated as:
  1. Very much improved
  2. much improved
  3. Minimally improved
  4. No change
  5. Minimally worse
  6. Much worse 7 = Very much worse
Time Frame: Visit 7: 52 weeks after baseline visit
Population: Eligible patients were older than 30 years; met the diagnostic criteria for possible or probable parkinsonism-predominant or cerebellar-ataxia-predominant multiple system atrophy; could ambulate independently (ie, Hoehn and Yahr stages 1-3); and had to be on stable anti-Parkinson's, anti-dysautonomia, anti-dementia, and anti-depressant regimens.
  In the EGCG group only 32 of 47 patients provided data at visit 5 due to SAE/drop out; likewise in the placebo group only 35 of 45 patients.
Measure: Number; unit: participants
Arm/Group | EGCG as Putative Neuroprotective Agent | Placebo
Number analyzed (Participants) | 32 | 35
participants
  global improvement =1 | 0 | 0
  global improvement =2 | 0 | 0
  global improvement =3 | 4 | 5
  global improvement =4 | 10 | 8
  global improvement =5 | 7 | 12
  global improvement =6 | 8 | 9
  global improvement =7 | 3 | 1

13. Secondary Outcome: Number of Participants Achieving Each Clinical Global Impression of Improvement (CGI-I): Efficacy Index (Therapeutic Effect of Treatment With Medication and Associated Side Effects) at Visit 7 Compared to the Baseline Visit
Description: The Clinical Global Impression - Efficacy Index is a 4×4 rating scale that assesses the therapeutic effect of treatment with psychiatric medication and associated side effects.
  It comprises 4 Items for the therapeutic effect:
  1. Marked - Vast improvement. Complete or nearly complete remission of all symptoms
  2. Moderate - Decided improvement. Partial remission of symptoms
  3. Minimal - Slight improvement which doesn't alter status of care of patient
  4. Unchanged or worse combined with 4 items of possible side effects: 1= None - no side effects (S.E.) 2= Side effects (S.E.) do not significantly interfere with patient's functioning 3= S.E. significantly interfere with patient's functioning 4= S. E. outweigh therapeutic effect The lowest total score (score 1) means vast improvement with no side effects; the highest total score (score 16) means unchanged or worse patient´s condition with side effects that outweigh the therapeutic effect.
Time Frame: Visit 7: 52 weeks after baseline visit
Population: Eligible patients were older than 30 years; met the diagnostic criteria for possible or probable parkinsonism-predominant or cerebellar-ataxia-predominant multiple system atrophy; could ambulate independently (ie, Hoehn and Yahr stages 1-3); and had to be on stable anti-Parkinson's, anti-dysautonomia, anti-dementia, and anti-depressant regimens.
  In the EGCG group only 32 of 47 patients provided data at visit 5 due to SAE/drop out; likewise in the placebo group only 30 of 45 patients.
Measure: Number; unit: participants
Arm/Group | EGCG as Putative Neuroprotective Agent | Placebo
Number analyzed (Participants) | 32 | 30
participants
  efficacy index score 5 (moderate therapeutic effect - no side effects | 0 | 1
  efficacy index score 7 (moderate therapeutic effect - side effects significantly interfering) | 1 | 0
  efficacy index score 9 (minimal therapeutic effect - no side effects | 1 | 1
  efficacy index score 11 (minimal therapeutic effect - side effects significantly interfering) | 0 | 1
  efficacy index score 13 (unchanged or worse -no side effects) | 28 | 26
  efficacy index score 14 (unchanged or worse -side effects not significantly interfering) | 1 | 0
  efficacy index score 15 (unchanged or worse -side effects significantly interfering) | 1 | 1

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: Adverse events were grouped according to Medical Dictionary for Regulatory Activities (MedDRA) organ class. Serious adverse events were defined as adverse events that led to hospitalisation, discontinuation of study medication because of liver toxicity, or death.
Arm/Group | EGCG as Putative Neuroprotective Agent | Placebo
All-Cause Mortality (participants affected / at risk) | 4/47 | 2/45
Serious Adverse Events (participants affected / at risk) | 18/47 | 8/45
Other Adverse Events (participants affected / at risk) | 25/47 | 33/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EGCG as Putative Neuroprotective Agent (N=47) | Placebo (N=45)
Hepatotoxicity (Hepatobiliary disorders) | 2 (2) | 0 (0) — Hepatotoxicity leading to discontinuation of study
Pneumonia due to aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Death (General disorders) | 4 (4) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
synkope (Cardiac disorders) | 1 (1) | 1 (1)
gastrointestinal disorders (Gastrointestinal disorders) | 5 (5) | 1 (1)
surgery (Surgical and medical procedures) | 1 (1) | 3 (3)
fracture of femoral bone (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
phlegmone hand (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
UTI (Renal and urinary disorders) | 0 (0) | 2 (2)
headache (Nervous system disorders) | 1 (1) | 0 (0)
heatstroke and exsikkosis (General disorders) | 1 (1) | 0 (0)
general worsening of overall health (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EGCG as Putative Neuroprotective Agent (N=47) | Placebo (N=45)
UTI (Renal and urinary disorders) | 9 (14) | 12 (18)
urinary dysfunction (Renal and urinary disorders) | 3 (3) | 6 (6)
dysarthria (Nervous system disorders) | 0 (0) | 4 (4)
dysphagia (Nervous system disorders) | 4 (5) | 0 (0)
falls (Nervous system disorders) | 17 (26) | 17 (31) — due to postural instability, ataxia or orthostatic hypotension
worsening of parkinsonism, ataxia or autonomic dysfunction (Nervous system disorders) | 10 (24) | 9 (17)
hepatotoxicity (Hepatobiliary disorders) | 6 (6) | 0 (0) — increased aminotransferase concentrations
orthostatic hypotension (Nervous system disorders) | 3 (6) | 5 (5)
gastrointestinal adverse event (Gastrointestinal disorders) | 17 (28) | 13 (21) — diarrhea, stomach pain, gastritis, constipation
swallowing problems (Nervous system disorders) | 3 (5) | 0 (0)
edema (Vascular disorders) | 3 (3) | 3 (3) — leg edema
depression (Psychiatric disorders) | 5 (5) | 2 (2)

LIMITATIONS AND CAVEATS:
The PROMESA trial had several limitations. The trial was powered to detect a 50% reduction in disease progression, not to detect smaller changes.

Furthermore, the assummed dropout rate was 20% while the observed drop out rate was approximately 27%. Furthermore, center size was heterogeneous, only four of the 12 centres recruited ten or more patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less